CLINICAL TRIAL: NCT00588653
Title: Diagnostic Accuracy of Capsule Endoscopy in Small Bowel Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Edward V. Loftus, Jr., M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2018-03
Record Dates: First submitted 2007-12-21; First posted 2008-01-08 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; capsule endoscopy; computed tomography enterography; colonoscopy; small bowel follow-through
MeSH Terms: conditions — Crohn Disease | interventions — Endoscopy; Colonoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): All patients were to undergo all 4 diagnostic modalities, and each of these was compared to the consensus clinical diagnosis. Readers of each modality were blinded to the results of the other 3.
  Interventions: Device: Capsule endoscopy, CT enterography, colonoscopy, small bowel follow-through

INTERVENTIONS:
Device: Capsule endoscopy, CT enterography, colonoscopy, small bowel follow-through — Each patient undergoes each of the 4 diagnostic modalities, but the readers are blinded to results of the other 3.

SUMMARY:
Prospective study to compare in a blinded fashion four different diagnostic modalities to detect active small bowel Crohn's disease: a) colonoscopy with ileoscopy; b) small bowel follow through; c) capsule endoscopy; and d) computed tomography enterography.

DETAILED DESCRIPTION:
Aims:

The aims of this study are as follows: 1) to describe the spectrum of small intestinal lesions demonstrated by capsule endoscopy (CE) in patients with Crohn's disease; 2) to determine the inter-observer agreement for recognizing these small intestinal lesions; 3) to determine the sensitivity, positive predictive value, and accuracy of CE, CT enterography, small bowel follow-through, colonoscopy with ileoscopy, and all pairwise combinations of these examinations with a consensus clinical diagnosis for the diagnosis and evaluation of the extent and severity of small intestinal Crohn's disease; 4) to establish a Crohn's Disease Capsule Endoscopy Index of Severity (CDCEIS); 5) to describe the spectrum of right colon lesions demonstrated by CE in patients with Crohn's disease.

Study Design and Methods:

Consecutive adult patients with suspected or definite Crohn's disease seen in the Inflammatory Bowel Disease Clinic at Mayo Clinic Rochester will be offered enrollment in a prospective observational trial comparing CE with CT enterography, small bowel follow-through, colonoscopy, and a consensus clinical diagnosis of Crohn's disease. Seventy patients will be enrolled, according to the inclusion and exclusion criteria, and written informed consent will be obtained. Co-investigators in the Inflammatory Bowel Disease (IBD) Clinic will clinically evaluate all patients, including a history and limited physical examination. Patients will undergo clinically indicated laboratory tests. Serum will be stored on all patients for other potential laboratory studies. Patients will complete a retrospective symptom diary for the week prior to their evaluation at Mayo, and a Crohn's Disease Activity Index (CDAI) will be calculated.

All patients will have a CT enterography with peroral contrast interpreted by a co-investigator radiologist. All patients will undergo a clinically indicated colonoscopy with ileoscopy by a staff co-investigator (not by C.A.S. or the staff co-investigator interpreting the CE), and a Crohn's Disease Endoscopic Index of Severity (CDEIS) will be calculated. If no significant small bowel strictures are identified by CT enterography or colonoscopy with ileoscopy, then patients will subsequently undergo CE. All CE studies will be read separately by C.A.S. (gastroenterology fellow) and a supervising staff gastroenterologist co-investigator, each blinded to the other's interpretation. The interobserver agreement between C.A.S. and the co-investigator staff will be determined. Patients will lastly have a clinically indicated small bowel follow-through interpreted by a co-investigator radiologist. All co-investigators will be blinded to the results of the other imaging modalities until after interpreting their respective studies.

Following each imaging procedure, the interpreting physician will complete both small intestine and colon anatomy forms. The physician will identify all types of lesions present and also give both a global evaluation of the severity of lesions found and a global Crohn's disease activity score indicating one of the following: active Crohn's disease, suspicious for Crohn's disease, inactive Crohn's disease, or no evidence of Crohn's disease. Co-investigators representing each of the diagnostic modalities will meet periodically to review those cases where there is disagreement among the imaging procedures with respect to the extent and severity of small intestinal Crohn's disease in order to reach a consensus clinical diagnosis. This consensus clinical diagnosis will serve as the gold standard against which each of the individual imaging modalities is evaluated. Sensitivity, positive predictive value, and accuracy of all diagnostic modalities compared to the consensus clinical diagnosis will be determined. A Crohn's disease capsule endoscopy index of severity (CDCEIS) will be created after the CE studies have been reviewed by investigators from other referral centers both inside and outside the United States to determine the inter-observer agreement (reproducibility) for each type of small bowel lesion identified by CE. Logistic regression analysis with step-wise deletion will then be utilized to create the CDCEIS using only those lesions that are reproducible, with the global Crohn's disease endoscopic activity score from the CE as the dependent variable.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient of either sex aged 18 to 70 years
* Patient has suspected or definite Crohn's disease
* Patient has read, understood, and signed a written informed consent form at visit 1.

Exclusion Criteria:

* Pregnancy
* Patients who are prisoners, institutionalized individuals, or vulnerable adults
* Patients immediately in need of abdominal surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, perforation, or intra-abdominal abscess
* Patients with known or suspected gastrointestinal obstruction due to significant stricture based upon the clinical symptoms (nausea, vomiting, abdominal distention, or abdominal pain) confirmed by pre-procedure evaluation. Pre-procedure evaluation includes CT enterography or small bowel follow through performed at Mayo or previously at an outside institution which demonstrates mechanical obstruction (mechanical obstruction defined as small bowel narrowing with pre-stenotic dilatation); additionally, a high-grade stenotic ileocecal valve or ileocolonic anastomosis found by colonoscopy.
* Patients with history of abdominal radiation
* Patients with known or suspected oropharyngeal or esophageal dysphagia (unless recent EGD shows no evidence of mechanical obstruction of the esophagus, in cases of esophageal dysphagia)
* Patients with pacemakers or other implantable electromedical devices
* Patients with highly suspected or documented gastroparesis
* Patients who have used NSAIDs within the previous 2 weeks
* Patients with an anticipated need for an MRI scan within two weeks after M2A capsule ingestion (for patients who require a clinically indicated MRI, the MRI should be performed prior to administration of the M2A capsule)
* Patients with a creatinine ≥ 2.0.
* Patients with documented reaction to iodinated contrast material.
* Patients with an ileostomy or colostomy
* Patients with documented reaction to metoclopramide.
* Patients with a hemoglobin less than 7.5 g/dl. (Patients with Crohn's disease are often chronically anemic, and a hemoglobin of 7.5 g/dl or greater would allow these patients to safely participate in the study.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-01; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity, positive predictive value, and accuracy of capsule endoscopy, CT enterography, colonoscopy with ileoscopy, and small bowel follow through using a consensus clinical diagnosis of small bowel Crohn's disease as the reference standard.

SECONDARY OUTCOMES:
Describe spectrum of right colon lesions visualized by capsule endoscopy in patients with Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Edward V Loftus, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States